CLINICAL TRIAL: NCT01291069
Title: Effect of Tadalafil on Exercise Capacity in Pediatric Fontan Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Shaji Menon, Assistant Professor, University of Utah
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB_00050085
Record Dates: First submitted 2011-02-04; First posted 2011-02-07 (Estimated); Last update posted 2017-04-17 (Actual); Status verified 2017-04

CONDITIONS: Single Ventricle
Keywords: Fontan; Tadalafil; Exercise performance
MeSH Terms: conditions — Univentricular Heart | interventions — Tadalafil; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tadalafil Citrate (Experimental): The study subjects will be given Tadalfil citrate, encapsulated, 0.8-1 mg/kg/day in 1 dose orally. Max dose 40 mg. All patients will receive either study drug or placebo for a total of 20 days.
  Interventions: Drug: Tadalafil Citrate
- Sugar pill (Placebo Comparator): If allocated to the placebo arm, the child will be given a similar appearing medication; the placebo will be a sugar pill. All patients will receive either study drug or placebo for a total of 20 days.
  Interventions: Drug: Sugar pill

INTERVENTIONS:
Drug: Tadalafil Citrate — If allocated to the treatment arm, the patient will be given tadalfil citrate, 0.8-1 mg/kg/day in 1 daily dose. Maximum dose 40 mg. All patients will receive either study drug or placebo for a total of 20 days.
  Other Names: Cialis
  Arms: Tadalafil Citrate
Drug: Sugar pill — If allocated to the placebo arm, the child will be given a similar appearing medication; the placebo will be a mixture of Ora-Sweet® and Ora-Plus® in a 1:1 ratio. All patients will receive drug for 20 days
  Other Names: Ora sweet
  Arms: Sugar pill

SUMMARY:
This pilot study is aimed at assessing the short-term effects of Tadalafil on the hemodynamic response to exercise and exercise capacity in patients with Fontan circulation. Data regarding effect size and drug tolerability will be used in the design of a randomized multicenter trial. The long-term goal of this investigation is to systematically evaluate the effect of tadalafil therapy on exercise performance, quality of life, and delay of functional deterioration in patients with single ventricle physiology.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have undergone the Fontan procedure (regardless of type of Fontan connection or presence or absence of a fenestration)
* Age 8.0 to 35.0 years
* Stable clinical condition over the last 3 months (i.e. No change in medication, treatments, or development of new symptoms)
* Ability to perform exercise testing
* Consent and assent (as appropriate to participate in the study after receiving information concerning procedures, risks, and possible clinical benefits) o Patients will be enrolled without regard to gender, race, and ethnicity. All patients meeting study eligibility will be approached for consent.

Exclusion Criteria:

* Severe heart failure (New York Heart Association functional class III or IV)
* Presence of liver or renal dysfunction based on the latest lab test results
* Presence of hearing or visual deficit
* Transcutaneous arterial blood oxygen saturation (SaO2) <80% at rest
* History of echocardiographic, MRI, or angiographic evidence of Fontan pathway obstruction
* History of exercise-induced life-threatening arrhythmias or unstable rhythm(i.e. atrial flutter)
* Known or suspected pregnancy. Females in the reproductive age group will be screened for pregnancy using serum beta hCG prior to administering study drug.
* Patients on open label sildenafil or tadalafil

Ages: 8 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2011-09; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
To compare the effects of Tadalafil versus placebo on exercise capacity (maximal oxygen consumption: VO2 max) for patients (8-35 years)with the Fontan circulation (8 -18 years). | 2 years
  Short-term treatment with Tadalafil will augment cardiac output and improve exercise capacity (maximal oxygen consumption: VO2 max) in patients with the Fontan circulation. Primary outcome variables include the change in peak exercise capacity (VO2 max), using cycle ergometry after one week of tadalafil therapy

SECONDARY OUTCOMES:
To evaluate the adverse effects of Tdalafil in patients (8-35 years)with the Fontan circulation and compare with the placebo group. | 2 years
  Hypothesis: Short-term treatment with Tadalafil will be well tolerated by children with the Fontan circulation. Adverse effect forms will be used to compare the side effects between Tadalafil and treatment group.

CONTACTS AND LOCATIONS:
Overall Officials: Shaji C. Menon, MD, Principal Investigator — University of Utah
Locations (1):
- Primary Childrens Medical Center, Salt Lake City, Utah, United States